CLINICAL TRIAL: NCT04910971
Title: Quantification of Binding and Neutralizing Antibody Levels in COVID-19 Vaccinated Health Care Workers Over 1 Year
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LifeBridge Health (Other)
Responsible Party: Principal Investigator, Paul A. Gurbel, Principal Investigator, LifeBridge Health
Other Study IDs: 1707882
Record Dates: First submitted 2021-06-01; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-06

CONDITIONS: COVID-19 Vaccine; Corona Virus Infection; Vaccine Adverse Reaction; Vaccine Response; Inflammation; Thrombosis
Keywords: Thrombosis; Inflammation; Vaccination; COVID-19
MeSH Terms: conditions — Coronavirus Infections; Inflammation; Thrombosis; COVID-19

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine for urinary 11-dehdro thromboxane Blood for platelet fibrin-clot strength as measured by Thrombelastography, IgG and IgM antibodies to SARS-CoV-2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Recipients of BNT162b2 mRNA Covid-19 Vaccine
- Group 2: Recipients of mRNA-1273 SARS-CoV-2 Vaccine

SUMMARY:
The severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) pandemic presents a great challenge to global health. The first case was identified in December 2019 in Wuhan, China and since has infected nearly 100 million people and claimed almost 2 million lives worldwide. In response, the medical community and scientists have worked hard to develop effective therapies and guidelines to treat a wide range of symptoms including the use of the antiviral drug remdesivir, convalescent plasma, antibiotics, steroids, and anticoagulant therapy. To prevent the spread of the disease, multiple vaccines based on mRNA and DNA technologies that include inactivated viral components have been developed and millions of doses are currently being administered worldwide. Early analysis of data from the phase III Pfizer/BioNTech and Moderna vaccine trials suggested the vaccine was more than 90% effective in preventing the illness with a good safety profile (Polack et al., 2020). However, there are still many unknowns regarding the long-term safety of these newer vaccine technologies and the level and duration of immunogenicity.

SARS-CoV-2 infection results in seroconversion and production of anti-SARS-CoV-2 antibodies. The antibodies may suppress viral replication through neutralization but might also participate in COVID-19 pathogenesis through a process termed antibody-dependent enhancement (Lu et al., 2020). Rapid progress has been made in the research of antibody response and therapy in COVID-19 patients, including characterization of the clinical features of antibody responses in different populations infected by SARS-CoV-2, treatment of COVID-19 patients with convalescent plasma and intravenous immunoglobin products, isolation and characterization of a large panel of monoclonal neutralizing antibodies and early clinical testing, as well as clinical results from several COVID-19 vaccine candidates.

In this study, we plan to assess the effic of both vaccines on the healthcare workers. As healthcare workers begin to receive their first vaccination dosage, we will start looking for traces of antibodies within the blood and saliva. The data provided will help us determine the efficacy of the vaccine over a period of 1 year, identify any difference in efficacy amongst different populations (gender, age, and ethnicities) differences among vaccine types, demographics and follow-up on any potential side effects. We will collaborate with Nirmidas Biotech Inc. based in Palto Alto, California, a Stanford University spinoff on this project. Nirmidas Biotech. Inc is a young diagnostic company that have received several FDA EUA tests for COVID-19. We will perform IgG/IgM antibody detection by the NIRMIDAS MidaSpot™ COVID-19 Antibody Combo Detection Kit approved by FDA EUA for POC testing in our hospital site for qualitative antibody testing. We will then send dry blood spot and saliva to Nirmidas for the pGOLD™ COVID-19 High Accuracy IgG/IgM Assay to quantify antibody levels and avidity, both of which are important to immunity. The pGOLD assay is a novel nanotechnology assay platform capable of quantifying antibody levels and binding affinity to viruses. We collaborated recently with Nirmidas on this platform and published a joint paper in Nature Biomedical Engineering on COVID-19 Ab pGOLD assay (Liu et al., 2020). It is also capable of detecting antibodies in saliva samples and could offer a non-invasive approach to assessing antibody response for vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females aged 18 years and older (inclusive) at screening.
* Able and willing (in the investigator's opinion) to comply with all study requirements.
* Willing to discuss their relevant medical history with the study investigators.
* Willing and able to give informed consent prior to study enrollment.

Exclusion Criteria:

* History of a recent or previous COVID-19 infection per history or as detected by either the PGOLD™COVID-19 IGG/IGM ASSAY or MidaSpot™ COVID-19 Antibody fingerstick test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health care workers within a large health care system being administered FDA approved SARS-CoV-2 vaccinations
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-01-31 (Actual); Primary Completion 2022-05-28 (Estimated); Study Completion 2022-07-28 (Estimated)

PRIMARY OUTCOMES:
Presence of IgG and IgM antibodies to SARS-CoV-2 in response to vaccination | 3 months
  Detection and quantification of IgG and IgM antibodies to SARS-CoV-2 by the antibody-avidity assay test
Loss of IgG and IgM antibodies to SARS-CoV-2 | 12 months
  Loss of IgG and IgM antibodies to SARS-CoV-2 when tested by the antibody-avidity assay test and rapid COVID-19 Antibody Combo Detection Kit at days 0, 20, 45, 70, 3 months, 6 months, 9 months, 12 months post-vaccination, after initial detection of antibodies

SECONDARY OUTCOMES:
Thrombo-inflammatory syndrome | 12 months
  Frequency of thrombo-inflammatory syndrome as defined by urinary 11-dehdro thromboxane > 4200 pg/mg in subjects experiencing a moderate-severe reaction to immunization
Side effects | 12 months
  he occurrence and severity of reactogenicity in terms of solicited local and systemic adverse events after each vaccination for the duration of 1 year.
Hypercoagulability | 12 months
  Frequency of hypercoagulability as defined by increased platelet fibrin-clot strength as measured by Thrombelastography in subjects experiencing a moderate-severe reaction to immunization

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Bliden, MBA, Study Director — Sinai Center for Thrombosis Research
Locations (1):
- Sinai Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No